CLINICAL TRIAL: NCT01025960
Title: Comparison of Detection of Polyps During Both Insertion and Withdrawal Phases of Colonoscopy Versus the Standard Practice of Detection of Polyps During the Withdrawal Phase of Colonoscopy: A Prospective Quality Improvement Study
Brief Title: A Comparison of Methods to Detect Polyps During Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 09-786
Record Dates: First submitted 2009-12-02; First posted 2009-12-04 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2012-03

CONDITIONS: Colorectal Cancer
Keywords: colonoscopy; adenoma detection; polyps
MeSH Terms: conditions — Colorectal Neoplasms; Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Inspection Colonoscopy (Other): The colonoscope will be inserted rapidly to reach the cecum. Inspection of the large bowel will occur during the withdrawal of the colonoscope.
  Interventions: Procedure: Standard Inspection Colonoscopy
- Dual Inspection Colonoscopy (Active Comparator): The large bowel will be inspected for polyps during the insertion of the colonoscope to the cecum, and during the withdrawal of the scope from the large bowel.
  Interventions: Procedure: Dual Inspection Colonoscopy

INTERVENTIONS:
Procedure: Standard Inspection Colonoscopy — The large bowel will be inspected for polyps during the withdrawal of the colonoscope to the cecum, and during the withdrawal of the scope from the large bowel.
  Arms: Standard Inspection Colonoscopy
Procedure: Dual Inspection Colonoscopy — The large bowel will be inspected for polyps during the insertion of the colonoscope to the cecum, and during the withdrawal of the scope from the large bowel.
  Arms: Dual Inspection Colonoscopy

SUMMARY:
Colorectal cancer (CRC) is the third most common cancer and second leading cause of cancer deaths in western countries. Colonoscopy is a preferred colorectal screening modality since it has both diagnostic and therapeutic capability. Detection and removal of polyps at colonoscopy decreases the incidence and mortality from colorectal cancer.

Typical practice is to insert the colonoscope rapidly until it reaches the cecum (a pouch-like portion of the intestines, where the large bowel and the small bowel meet). The physician then withdraws the colonoscope slowly and looks for any polyps or abnormalities within the large bowel. The purpose of this study is to compare this standard practice to the approach whereby the physician examines the bowel as the scope is initially inserted AND as the colonoscope is withdrawn from patients' colons.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Patients able to provide an informed consent
* Patients undergoing colonoscopy

Exclusion Criteria:

* Pregnant women
* Patients with Familial Adenomatous Polyposis Syndromes (FAP)
* Patients with Hereditary Non-polyposis Colon Cancer Syndrome (HNPCC)
* Patients who have undergone previous surgical resection of the colon
* Patients who have been diagnosed with inflammatory bowel disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 768 (Actual)
Dates: Start 2009-11; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Adenoma detection rates for each method | within the first 30 days after colonoscopy

SECONDARY OUTCOMES:
Comparison of procedure times for each method | 1 year
Percentage of patients with at least one adenoma detected by each method | 1 year
Comparison of percentage of adenomas classified as high risk for each method | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Madhusudhan Sanaka, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Sanaka MR, Parsi MA, Burke CA, Barnes D, Church J, Rizk M, Zein N, Joseph R, Thota PN, Lopez R, Kiran RP. Adenoma detection at colonoscopy by polypectomy in withdrawal only versus both insertion and withdrawal: a randomized controlled trial. Surg Endosc. 2015 Mar;29(3):692-9. doi: 10.1007/s00464-014-3723-3. Epub 2014 Jul 19. PMID 25037727